CLINICAL TRIAL: NCT04427189
Title: Better Control in Pediatric and Adolescent diabeteS: Working to crEate CEnTers of Reference
Brief Title: Better Control in Pediatric and Adolescent diabeteS: Working to crEate CEnTers of Reference (SWEET- Registry)
Acronym: SWEET
Status: Recruiting | Type: Observational
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Collaborators: SWEET e.V (Unknown)
Responsible Party: Principal Investigator, Olga Kordonouri, Prof. Dr., Kinderkrankenhaus auf der Bult
Other Study IDs: SWEET-10
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes
Keywords: Pediatric
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SWEET-REGISTRY is a multi center, investigator initiated registry in patients with diabetes. SWEET' is an acronym derived from 'Better control in Pediatric and Adolescent diabeteS: Working to crEate CEnTers of Reference'. Having the vision of equal quality care for all children with diabetes the mission of SWEET is to harmonize care to optimize outcomes of children with diabetes worldwide. Initiated with support of the EU Public Health Program in 2008 the SWEET group has over 10 years of experience in creating and sustaining a high quality professional network based on agreed standards of care, criteria for certification, international guidelines and quality control. While originally focusing on the European region, SWEET is currently expanding and has received increasingly global attention, with centers across different continents including Asia, Africa, North and South-America. SWEET extracts wherever possible the data from existing data collection sources and following longitudinally unselected clinical populations of all pediatric diabetes patients as an ongoing measure of benchmarking and a quality control cycle as well as a resource for scientific studies and collaborative research. The SWEET registry was approved by the ethical committee of Hannover Medical School and is associated with the AUF DER BULT Diabetes Centre for Children and Adolescents, Hannover, Germany, which coordinates the SWEET collaboration. Each center has to meet specific entry criteria showing diabetes expertise and compliance with the International Society for Pediatric and Adolescent Diabetes (ISPAD) clinical practice guidelines. The local institutional review boards of the participating centers approved the pseudonymized data collection.

DETAILED DESCRIPTION:
The SWEET-Registry is a prospective evaluation of the effectiveness of multidisciplinary treatment approaches of international pediatric diabetes centers.The hypothesis is that a collaboration of pediatric diabetes centers will improve the situation for children with diabetes ensuring that all children have the right to participate fully in all the experiences of childhood and adolescence, regardless of whether they have diabetes and wherever they live. Also it could reduce the effects of accelerated vascular ageing imposed by the diabetic state and provide the basis for a long-term participation in professional and family life without or with delayed debilitating long-term diabetes complications.

SWEET is a real-world study. Therefore the treatment decisions are made by the patient with diabetes and the local treatment team.

The SWEET database combines data from distinct sources. Data is collected locally through clinical databases, electronic health record systems, the standardized SWEET-DPV-documentation software (https://sweet.zibmt.uni-ulm.de/software.php) or centers download data from existing longitudinal registries. Twice yearly, data are transmitted to the central database hosted by the Institute of Epidemiology and Medical Biometry, ZIBMT, Ulm University, Ulm, Germany. The prospectively collected data is then combined into a common database. Inconsistent/improbability or missing data is reported back to the centers for correction. Data is then aggregated into an anonymized, cumulative database used for clinical research, scientific analysis, and nationwide benchmarking.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus (as diagnosed clinically)
2. Males and females of all Ages, but with a focus on pediatric care
3. Provision of informed consent from participant and all legal representatives prior to any study specific procedures

Exclusion Criteria:

1. no diabetes
2. no consent,
3. Patient who, in the judgment of the Investigator, is found to be unlikely to comply with the protocol, or has any severe concurrent medical or psychological condition that may affect the interpretation of efficacy or safety data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from Diabetes centres worldwide diagnosed with Diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2008-04 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change of HbA1c level | through study completion, an average of 1 year, up to 5 years
  assessment of the metabolic situation based on the level of HbA1c

SECONDARY OUTCOMES:
hypoglycemia rate | through study completion, an average of 1 year, up to 5 years
  number of events of severe hypoglycemia
Time in Range | through study completion, an average of 1 year, up to 5 years
  percentage of CGM values between 70-180 mg/dl
DKA rate | through study completion, an average of 1 year, up to 5 years
  number of hospitalizations due to DKA

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Danne, MD, Principal Investigator — Kinderkrankenhaus auf der Bult
Locations (1):
- Kinderkrankenhaus auf der Bult, Hanover, Low Saxony, Germany

REFERENCES:
- [Derived] Chobot A, Eckert AJ, Biester T, Corathers S, Covinhas A, de Beaufort C, Imane Z, Kim J, Malatynska A, Moravej H, Pokhrel S, Skinner T, Study Group S. Psychological Care for Children and Adolescents with Diabetes and Patient Outcomes: Results from the International Pediatric Registry SWEET. Pediatr Diabetes. 2023 Jun 2;2023:8578231. doi: 10.1155/2023/8578231. eCollection 2023. PMID 40303253
- [Derived] Limbert C, Lanzinger S, deBeaufort C, Iotova V, Pelicand J, Prieto M, Schiaffini R, Sumnik Z, Pacaud D; SWEET Study Group. Diabetes-related antibody-testing is a valuable screening tool for identifying monogenic diabetes - A survey from the worldwide SWEET registry. Diabetes Res Clin Pract. 2022 Oct;192:110110. doi: 10.1016/j.diabres.2022.110110. Epub 2022 Sep 30. PMID 36183869
- [Derived] Danne T, Lanzinger S, de Bock M, Rhodes ET, Alonso GT, Barat P, Elhenawy Y, Kershaw M, Saboo B, Scharf Pinto M, Chobot A, Dovc K. A Worldwide Perspective on COVID-19 and Diabetes Management in 22,820 Children from the SWEET Project: Diabetic Ketoacidosis Rates Increase and Glycemic Control Is Maintained. Diabetes Technol Ther. 2021 Sep;23(9):632-641. doi: 10.1089/dia.2021.0110. Epub 2021 Aug 18. PMID 34086503
- [Derived] Gerhardsson P, Schwandt A, Witsch M, Kordonouri O, Svensson J, Forsander G, Battelino T, Veeze H, Danne T. The SWEET Project 10-Year Benchmarking in 19 Countries Worldwide Is Associated with Improved HbA1c and Increased Use of Diabetes Technology in Youth with Type 1 Diabetes. Diabetes Technol Ther. 2021 Jul;23(7):491-499. doi: 10.1089/dia.2020.0618. Epub 2021 Feb 26. PMID 33566729